CLINICAL TRIAL: NCT07206667
Title: Improved Understanding of Venous Drainage at the Cranio-cervical Junction : Study of Postoperative Venous Remodeling Following Surgical Treatment of Lesions of the Posterior Fossa or Posterior Approach of the Upper Cervical Spine.
Acronym: VENAMAP 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC24.0305; 2025-A00646-43 (Other: ANSM)
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Craniocervical Surgery
Keywords: neurosurgery; cerebral venous drainage; MRI

STUDY DESIGN:
Intervention Model Description: Single-center exploratory prospective study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (all patients) (Experimental): During the two routine MRI scans, a T1 GRE GADO MRI sequence (specific to the study) will be added. It lasts approximately 3 minutes.
  Interventions: Procedure: T1 GRE GADO MRI sequence

INTERVENTIONS:
Procedure: T1 GRE GADO MRI sequence — Addition of a T1 gradient echo sequence with gadolinium (T1 TFE GADO) during the two MRI scans performed in routine practice before and after neurosurgery.

SUMMARY:
In the literature, we most often find a dichotomous view of cerebral venous drainage. Thus, two drainage pathways are most often considered: the jugular vein network and the vertebral artery plexus. However, several clinical observations seem to indicate a much more complex situation.

The following hypothesis is therefore put forward: there are alternative drainage pathways to these main pathways, which are physiologically present and capable of draining a significant volume of blood. A set of alternative pathways, which can be described as "deep," has been described: in particular, drainage pathways surrounding the vertebral artery (vertebral artery venous plexus), epidural plexuses, and deep cervical veins. However, the so-called "superficial" systems (subcutaneous and muscular) do not appear to have been studied.

There appears to be a change in venous drainage of the craniocervical junction postoperatively (posterior cranial fossa surgery and posterior approach to the upper cervical spine).

These modifications would vary depending on the venous drainage configuration present in each patient. If this hypothesis is confirmed, it could have an impact on the management of each patient. Thus, if venous remodeling models are established, this could enable personalized perioperative patient management: better optimization of body position during installation in the operating room, more effective anticipation of potential intraoperative venous bleeding, and explanation of persistent headaches in the postoperative period due to insufficient compensation of venous drainage. Confirmation of this hypothesis would also improve our understanding of certain pathologies for which the venous hypothesis has been raised (chronic hydrocephalus in adults, idiopathic intracranial hypertension, etc.).

DETAILED DESCRIPTION:
Inclusion:

The inclusion visit will take place during an initial neurosurgery consultation. If the patient meets the inclusion and exclusion criteria and wishes to participate in this study, the study investigator will obtain the patient's consent.

During this visit, a routine MRI will be performed if the patient has not already had one. In addition to the standard procedure, this MRI will include the study-specific T1 GRE GADO MRI sequence, which will add approximately 3 minutes to the usual examination. The patient will also undergo a routine neurological clinical examination and data about them will be collected (informative data about the patient (age, sex, BMI, etc.), medical history, neurological functional signs, reason for treatment, and neurological clinical examination).

First follow-up visit:

During hospitalization in the neurosurgery department, the patient will undergo a routine neurological clinical examination and data will be collected intraoperatively (duration of surgery, blood loss, ligation/clipping/any interventions on venous structures, intraoperative hemorrhage, other complications of all types) as well as early postoperative data (complications, types, headaches).

The time between the preoperative visit and surgery varies and may depend on the patient's surgical indication.

Second follow-up visit:

Finally, the patient will be asked to come to the neurosurgery department for a post-operative visit a few weeks after their surgery.

This visit is part of standard practice and includes a clinical neurological examination.

During this visit, a second MRI will be performed using the specific sequence for the study, T1 GRE GADO, which will add approximately 3 minutes to the routine examination. Data concerning the patient will be collected (complications, types, headaches).

ELIGIBILITY:
Inclusion Criteria:

Patient:

* Adult
* Surgery of the posterior cranial fossa or posterior approach to the upper cervical spine, regardless of indication, performed in the neurosurgery department at Brest University Hospital
* Having undergone an MRI with T1 echo gradient sequence with gadolinium (T1 TFE GADO)
* Affiliated with a Social Security scheme
* Having given written consent to participate in the study

Exclusion Criteria:

* Pregnant or breastfeeding women
* Allergy to gadolinium
* Any contraindications to undergoing an MRI scan (incompatible medical device implant, claustrophobia, etc.)
* Patients unable to understand the protocol
* Patients under guardianship or conservatorship
* Patients subject to a future protection order, family authorization, or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Dominant network before and after surgery in the craniocervical junction | Pre-surgery MRI (performed up to 12 weeks before surgery) + Post-surgery MRI (performed between 10 days and 16 weeks after surgery)
  The primary endpoint is identification of the dominant network before and after surgery in the craniocervical junction (i.e., 3 months after surgery).
  A T1 echo gradient sequence with gadolinium (T1 TFE GADO), lasting approximately 3 minutes, will be added to the MRIs performed as part of routine care before and after surgery on patients.
  A double reading of the MRI will be performed:
  * First by a neurosurgery intern,
  * Secondly, by a senior neuroradiology investigator who is blinded to the measurements taken by the neurosurgery intern.
  * In the event of a discrepancy between the two observers, the values obtained by the senior radiologist will be retained.
  The percentage change in the dominant network will be presented with its 95% confidence interval.

SECONDARY OUTCOMES:
Dominant network before and after surgery in the craniocervical junction and type of surgery | Pre-surgery MRI (performed up to 12 weeks before surgery) + Post-surgery MRI (performed between 10 days and 16 weeks after surgery)
  A T1 echo gradient sequence with gadolinium (T1 TFE GADO), lasting approximately 3 minutes, will be added to the MRIs performed as part of routine care before and after surgery on patients.
  A double reading of the MRI will be performed:
  * First by a neurosurgery intern,
  * Secondly, by a senior neuroradiology investigator who is blinded to the measurements taken by the neurosurgery intern.
  * In the event of a discrepancy between the two observers, the values obtained by the senior radiologist will be retained.
  The percentage change in dominant network by type of surgery (Oncological skull surgery, Non-oncological skull surgery, Emergency spinal surgery and Elective spinal surgery) and the percentage change in lateralization of dominance will be presented with their 95% confidence interval.
Dominance (right/left) of venous drainage before and after surgery | Pre-surgery MRI (performed up to 12 weeks before surgery) + Post-surgery MRI (performed between 10 days and 16 weeks after surgery)
  A T1 echo gradient sequence with gadolinium (T1 TFE GADO), lasting approximately 3 minutes, will be added to the MRIs performed as part of routine care before and after surgery on patients.
  A double reading of the MRI will be performed:
  * First by a neurosurgery intern,
  * Secondly, by a senior neuroradiology investigator who is blinded to the measurements taken by the neurosurgery intern.
  * In the event of a discrepancy between the two observers, the values obtained by the senior radiologist will be retained.
  The percentage change in dominant network by type of surgery and the percentage change in lateralization of dominance will be presented with their 95% confidence interval.
Total surface area of vessels before and after surgery, overall and within each venous network of the craniocervical junction. | Pre-surgery MRI (performed up to 12 weeks before surgery) + Post-surgery MRI (performed between 10 days and 16 weeks after surgery)
  A T1 echo gradient sequence with gadolinium (T1 TFE GADO), lasting approximately 3 minutes, will be added to the MRIs performed as part of routine care before and after surgery on patients.
  A double reading of the MRI will be performed:
  * First by a neurosurgery intern,
  * Secondly, by a senior neuroradiology investigator who is blinded to the measurements taken by the neurosurgery intern.
  * In the event of a discrepancy between the two observers, the values obtained by the senior radiologist will be retained.
  The mean surface differences (overall, by venous network, and by lateralization of initial dominance) will be presented with their 95% confidence interval.
Total surface area of vessels before and after surgery and initial dominance | Pre-surgery MRI (performed up to 12 weeks before surgery) + Post-surgery MRI (performed between 10 days and 16 weeks after surgery)
  A T1 echo gradient sequence with gadolinium (T1 TFE GADO), lasting approximately 3 minutes, will be added to the MRIs performed as part of routine care before and after surgery on patients.
  A double reading of the MRI will be performed:
  * First by a neurosurgery intern,
  * Secondly, by a senior neuroradiology investigator who is blinded to the measurements taken by the neurosurgery intern.
  * In the event of a discrepancy between the two observers, the values obtained by the senior radiologist will be retained.
  The mean surface differences (overall, by venous network, and by lateralization of initial dominance) will be presented with their 95% confidence interval.
Vessel diameter according to internal assessment and senior radiologist | Pre-surgery MRI (performed up to 12 weeks before surgery) + Post-surgery MRI (performed between 10 days and 16 weeks after surgery)
  The agreement between the measurement of vessel diameters by the intern or the experienced radiologist will be assessed graphically using the Bland and Altman method and numerically using the intraclass correlation coefficient accompanied by its 95% confidence interval estimated using the Fleiss method. The intraclass correlation coefficient will be interpreted using the following correspondences:
  * < 0.50: Unacceptable
  * 0.51-0.60: Low
  * 0.61-0.70: Mediocre
  * 0.71-0.80: Satisfactory
  * 0.81-0.90: Fairly good
  * 0.91-0.95: Very good
  * 0.95: Excellent

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, Brittany Region, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.